CLINICAL TRIAL: NCT03266679
Title: Bipolar Mood Disorders: A Recovery-Oriented Intervention Approach Addressing Deficits In Metacognitive Capacities
Brief Title: Psychological Factors In The Treatment Of Bipolar Mood Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queensland University of Technology (Other)
Collaborators: Metro South Health Addiction & Mental Health Services (Unknown)
Responsible Party: Principal Investigator, Priyanka Komandur, PhD Student/Clinical Psychology Registrar, Queensland University of Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ethics Approval No: 1700000591
Record Dates: First submitted 2017-08-13; First posted 2017-08-30 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Metacognitive Capacities
Keywords: bipolar disorder; metacognition; reflective functioning; metacognition-based intervention; sense of self; insight
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Intervention Model Description: Case-Series Design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients receiving metacognition-based intervention (Other): Case-Series Design - all participants receive the intervention - metacognition-based therapy (adapted version of Metacognitive Reflection and Insight Therapy developed by Lysaker & Klion) - weekly for a period of 12 months. No control/comparison group.
  Interventions: Other: Metacognitive Reflection and Insight Therapy - Adapted

INTERVENTIONS:
Other: Metacognitive Reflection and Insight Therapy - Adapted — The intervention involves the following elements: setting an agenda, developing a therapeutic relationship, therapist transparency and insertion of therapist's mind, analysis of narrative episodes, problem definition, stimulating self-reflection and understanding of others, stimulating mastery, reflecting on therapeutic relationship, and client assessment of outcomes.

SUMMARY:
The aim of this study is to trial an intervention targeting potential deficits in an individual's ability to form, and reflect upon, ideas about themselves and others (known as metacognitive capacities), specifically in relation to individuals diagnosed with a bipolar mood disorder (BMD).

The proposed research will adopt a mixed qualitative and quantitative design. Participants will be recruited through hospital outpatient groups (i.e., Metro South Addiction & Mental Health Services Woolloongabba Community Health Centre & Beenleigh Community Health Centre in Brisbane, Queensland), and, as necessary, local non government organisations (NGOs), psychiatrists, general practitioners, online support networks (SANE Australia, Black Dog Institute), community mental health services(such as MINDNET), and/or social media groups (Facebook, Twitter) supporting people who meet criteria for a BMD. The research will then use clinical interviews and quantitative (survey) methods to: (1) confirm diagnosis of participants; and (2) confirm deficits in metacognitive capacities of participants. Following this, the research will then involve the implementation of an adapted intervention across a course of 12 months, aimed at improving the metacognitive capacities of participants with a diagnosis of a BMD.

The research will provide an enriched understanding of a dimension of people with BMDs that has not been previously explored. The research will help with gaining an understanding of the metacognitive processes of people with BMDs, and inform more targeted psychological interventions.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with a Bipolar Affective (mood) Disorder
* Medication has not been changed for at least the past one month
* No hospitalisations in the past month
* Able to provide informed consent

Exclusion Criteria:

* Diagnosed with an Intellectual Disability
* Diagnosed with Schizoaffective Disorder
* High risk of suicide; defined as current, daily suicidal ideation, or the presence of a current plan and intent to commit suicide

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-07-26 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
The Indiana Psychiatric Illness Interview (IPII) | IPII + MAS-A (see below) combined take approximately 45- 60 minutes
  The IPII is a semi-structured interview that will be used to assess how participants understand their experience with mental illness (i.e., to elicit and assess an illness narrative). The interview is conceptually divided into five sections. First, rapport is established and participants are asked to tell the story of their lives, beginning with their earliest memory. Second, participants are asked if they think they have a mental illness and, if so, whether or not this condition has affected different facets of their life. Third, participants are asked if and how their condition controls their life and, alternately, how they control their condition. Fourth, they are asked how their condition affects, and is affected by others. Finally, participants are asked about their expectations for the future. The narratives of self and illness are then qualitatively analysed (form and quality rather than content) and then quantitatively rated.
The Metacognition Assessment Scale - Abbreviated (MAS-A) | IPII + MAS-A combined take approximately 45-60 minutes
  The MAS-A is an observer rating scale that will be used to assess metacognitive capacity. The MAS-A can be used either in a structured interview format or during a therapy session. The measure presumes that metacognition is comprised of multiple related but semi-independent functions. The MAS-A provides an overall measure of metacognitive capacity, as well as four subscale measures. The four subscales are: 1) Self-reflectivity or Understanding of One's Own Mind - the ability of a person to think about his or her own mental states; 2) Understanding Others' Minds - the ability to think about the mental states of others; 3) Decentration - the ability to see other's mental states with motivations and hypotheses independent from their own); and, 4) Mastery - the ability to use
The Narrative Coherence Rating Scale (NCRS) | 10-15 minutes
  The NCRS is a six item, 18-point rating scale developed to assess narrative coherence of illness narratives elicited from the IPII. The six items are: 1) "Logical connections" among the narrative of past psychiatric illnesses; 2) "Logical connections" among the narrative of psychiatric illnesses in the present; 3) "Richness of historical detail" among the narrative of past psychiatric illnesses; 4) "Richness of historical detail" among the narrative of psychiatric illnesses in the present; 5) "Plausibility" among the narrative of psychiatric illnesses in the past; and 6) "Plausibility" among the narrative of psychiatric illnesses in the present. A trained rater reviews an IPII transcript and rates according to scoring anchors (Lysaker et al., 2002).

SECONDARY OUTCOMES:
Treatment Outcome Package (TOP) | 15-20 minutes
  The TOP is a multidimensional outcome measure designed to track behavioural health treatment progress and outcomes. The TOP has three age-specific versions (child, adolescent, adult). The adult TOP clinical scales consist of 58 items assessing 12 symptom and functional domains: work functioning, sexual functioning, social conflict, depression, panic (somatic anxiety), psychosis, suicidal ideation, violence, mania, sleep, substance abuse, and quality of life. Items (e.g., "Felt down or depressed" "Felt on top of the world") can be summed across the domains to form a global symptom severity score. When using raw (non-standardised) scores, higher TOP total scores indicate healthier functioning. The TOP clinical scales and total score have demonstrated adequate internal consistency reliability and test-retest reliability, and convergent, discriminant, and criterion validity (Kraus, Seligman, & Jordan, 2005).
The Hamilton Depression Rating Scale (HDRS) | 10 minutes
  The HDRS is a 17-item, clinician-rated scale that will be used to assess the severity of, and change in, depressive symptoms in participants over the past week. Items (e.g., Feelings of Guilt) are rated on scales of varying grades of severity (e.g., 0 = absent, 4 = incapacitating). The HDRS item scores can be summed to obtain a total score (ranging from 0 to 52), where higher scores indicate greater depression severity. The HDRS has demonstrated adequate reliability (internal, interrater, and retest) and validity (convergent, discriminant, and predictive; Bagby, Ryder, Schuller, Marshall, 2004).
The Young Mania Rating Scale (YMRS) | 10 minutes
  The YMRS is an 11-item, clinician-rated scale that will be used to assess symptoms of mania over the past week. There are four items (Irritability, Speech, Thought Content, and Disruptive/Aggressive Behaviour) that are rated on a 0 to 8 scale, while the remaining items are rated on a 0 to 4 scale. All rating scales have explicitly described grades of severity. The YMRS scores can be summed to obtain a total score (ranging from 0 to 60), where higher scores indicate greater severity of the symptom. The YMRS has demonstrated adequate internal consistency and test-retest reliability, as well as convergent and divergent validity (Young et al., 1978).
The Sheehan Disability Scale (SDS) | 1-2 minutes
  The SDS is a 5-item, self-reported questionnaire used to measure the extent to which an individual's disability due to an illness or health problem has interfered with: (1) work/school; (2) social life/leisure activities (3) and family life/home responsibilities (each area is considered a subscale of the questionnaire) in the past week. The first three items (e.g.,"The symptoms have disrupted your work/school work") are rated on a Likert-type scale (0 = not at all, 10 = extremely). Each subscale can be scored separately or combined into a total score (sum of non-missing responses) ranging from 0 to 30, where higher scores indicate significant functional impairment.
The 36-Item Short Form Healthy Survey (SF-36) | 5-10 minutes
  The SF-36 is a 36-item scale used to measure an individual's QoL. The scale taps into varying health concepts, with eight subscales: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. It also includes a single item that provides an indication of perceived change in health. Items (e.g., "How much bodily pain have you had in the past 4 weeks?") are rated on Likert-type scales of varying ranges (between 1-2 and 1-6). Items in the same scale are averaged together to form eight scale scores (average is based on questions that received a response, missing data is excluded). Items are scored such that higher scores indicate a more favourable health state (Ware Jr & Sherbourne, 1992).
The Inventory of Interpersonal Difficulties (IIP-32) | 5 minutes
  The IIP-32 is a 32-item self-report questionnaire used to measure the severity of a wide range of difficulties experienced in interpersonal relationships. It is a shortened version of the 127-item IIP (Horowitz, Rosenberg, Baer, Ureno, & Villasenor, 1998) The scale comprises eight subscales: hard to be sociable, hard to be assertive, too aggressive, too open, too caring, hard to be supportive, hard to be involved, and too dependent. Items (e.g., "I open up to people too much") are rated on a 5-point Likert-type scale ranging from 0 (not at all) to 4 (extremely), where higher scores indicate greater severity of difficulties experienced. Correlations between the mean item score on the IIP and the IIP-32 were .94 and .96, respectively, at pre- and post-treatment administrations in an efficacy study of time-limited treatment for depression (Barkham, Hardy, & Startup, 1996).

CONTACTS AND LOCATIONS:
Overall Officials: Priyanka Komandur, Principal Investigator — Queensland University of Technology
Locations (2):
- Australia (2):
  - Queensland University of Technology, Brisbane, Queensland
  - Metro South Addiction & Mental Health Services, Brisbane, Queensland

IPD SHARING:
Plan to Share IPD: No